CLINICAL TRIAL: NCT04251442
Title: Randomized Controlled Trial of Patients Undergoing a Total Knee Arthroplasty With and Without the Use of Intraoperative Sensing Technology
Brief Title: TKR With and Without the Use of Intra-operative Sensing
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Per funding institution
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Orthosensor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-0144
Record Dates: First submitted 2020-01-29; First posted 2020-02-05 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Total knee repalcement
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Study Group (Experimental): The study group will have soft tissue balance performed with the use of IOS.
  Interventions: Device: OrthoSensor Verasense Technology
- Control Group (No Intervention): Control group patients will have soft tissue balance performed manually, with final soft tissue balance values measured using IOS, while the surgeon will remain blinded to those values.

INTERVENTIONS:
Device: OrthoSensor Verasense Technology — IOS is used to send real time information to a monitor within the operating room that assists your surgeon in making decisions about the balance of the ligaments in your knee and the proper insertion of implants.
  Arms: Study Group

SUMMARY:
The purpose of this study is to determine if there is a difference in clinical outcomes after total knee replacement (TKR) performed with traditional ligament balancing compared to use of intraoperative sensing technology (IOS) to balance ligaments. IOS is used to send real time information to a monitor within the operating room that assists your surgeon in making decisions about the balance of the ligaments in your knee and the proper insertion of implants. A total of 150 subjects will participate in this study at Hospital for Special Surgery.

The hypotheses are that the use of IOS technology will be associated with:

1. Better soft tissue balance during TKR than by manual balancing alone.
2. Higher patient reported clinical outcome measures (PROMs) following surgery.

DETAILED DESCRIPTION:
Participation in this study will involve a knee replacement performed with IOS. Patients will be randomized into one of two groups:The study group will have soft tissue balance performed with the use of IOS. Control group patients will have soft tissue balance performed manually, with final soft tissue balance values measured using IOS, while the surgeon will remain blinded to those values. Intra-operative compartment loads will be measured in 10, 45, and 90 degrees of flexion.

Additionally, long leg limb alignment, passive range of motion, use of opioids, daily activity, and PROMS will be evaluated post-operatively to determine which group has better outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet the indications for use for primary TKR using IOS
* Subject must be diagnosed with osteoarthritis
* Subject is likely to be available for all study visits
* Subject is able and willing to sign the informed consent and follow study procedures

Exclusion Criteria:

* Revision total knee arthroplasty
* Patient is receiving treatment for any of the following conditions:

  1. Avascular Necrosis
  2. Inflammatory arthritis
  3. Post-traumatic arthritis
* Any knee surgery other than meniscectomy (can be arthroscopic or open)
* Ligament insufficiencies, prior surgeries such as anterior cruciate ligament (ACL) or posterior cruciate ligament (PCL) reconstructions, posterolateral reconstructions, osteotomies, tibia plateau fractures
* Ipsilateral foot/ankle and hip arthritis
* Range of motion less than 90°
* Subject has a mental condition that may interfere with the subject's ability to give an informed consent or willingness to fulfill the study requirements (i.e. severe mental retardation such that the Subject cannot understand the informed consent process, global dementia, prior strokes that interfere with the Subject's cognitive abilities, senile dementia, and Alzheimer's Disease)
* Any subjects meeting any contraindication criteria as identified in the locally approved labeling for the device should be excluded from this study.
* Patient out-of-state with medication prescription not registered in iStop database
* Patients with severe contralateral osteoarthritis requiring subsequent knee replacement or with a flexion contracture greater than 10 degrees.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Knee Society Score | 4 months
  The primary outcome will be the difference in Knee Society Score (KSS) between baseline and 4 months post-operatively. The Knee Society Score is out of 100 points, with a higher score meaning a patient had a better outcome.

SECONDARY OUTCOMES:
Intra-operative Compartment Loads | Intra-operative
  Intra-operative compartment loads (medial and lateral component loads) will be measured between the groups at 10, 45, and 90 degrees of flexion during trial reduction and after cementation, using IOS technology.
Long Leg Limb Alignment | 6 weeks
  Long leg limb alignment will be measured on post-operative standard of care (SOC) radiographs at patients' 6 week follow-ups.
Passive Range of Motion | 4 months
  Passive range of motion will be measured pre-operatively, 6 weeks post-operatively, and 4 months post-operatively at all scheduled SOC appointments.
Opioid Use | 6 weeks
  Use of opioids will be tracked using the Internet System for Tracking Over Prescribing (I-STOP) database and a daily pain diary maintained by patient for first 6 weeks post-operatively. The I-STOP database can be accessed by the prescribing physician to track how many opioid refills a patient has procured.
Function and Activity | 6 weeks
  Function and activity will be monitored using Fitness Trackers. The device will be given to each patient in hospital and is to be worn for 6 weeks post-operatively. It will monitor a patient's daily and weekly steps while the patient is wearing it.
Pain Level | 6 weeks
  Daily pain levels will also be measured using the fitness tracker. The tracker will ask the patient to rate their pain on a scale from 0-10, with 0 meaning they have no pain, and 10 being the worst pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Gonzalez Della Valle, MD, Principal Investigator — Hospital for Special Surgery, New York; Kate Shanaghan, Study Director — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cho KJ, Seon JK, Jang WY, Park CG, Song EK. Objective quantification of ligament balancing using VERASENSE in measured resection and modified gap balance total knee arthroplasty. BMC Musculoskelet Disord. 2018 Jul 27;19(1):266. doi: 10.1186/s12891-018-2190-8. PMID 30053812
- [Result] Nodzo SR, Franceschini V, Gonzalez Della Valle A. Intraoperative Load-Sensing Variability During Cemented, Posterior-Stabilized Total Knee Arthroplasty. J Arthroplasty. 2017 Jan;32(1):66-70. doi: 10.1016/j.arth.2016.06.029. Epub 2016 Jun 22. PMID 27436499